CLINICAL TRIAL: NCT03333499
Title: the Effects of YangXinShi (YXS) on the Quality of Life and Exercise Tolerance in Patients With Chronic Heart Failure
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dalian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: zsyy_xhs2017-10
Record Dates: First submitted 2017-10-20; First posted 2017-11-07 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- the control group (Placebo Comparator): YanXinShi placebo pills
  Interventions: Drug: YanXinShi placebo pills
- YanXinShi group (Experimental): YanXinShi pills
  Interventions: Drug: YanXinShi pills
- Trimetazidine group (Active Comparator): Trimetazidine pills
  Interventions: Drug: Trimetazidine pills
- YangXinShi and Trimetazidine group (Other): YanXinShi and Trimetazidine pills
  Interventions: Drug: YanXinShi and Trimetazidine pills

INTERVENTIONS:
Drug: YanXinShi placebo pills — participants will take matched 1800 mg YXS placebo pills TID in addition to the optimal combination drug treatment of heart failure
  Arms: the control group
Drug: YanXinShi pills — participants will take 1800 mg YXS pills TID in addition to the optimal combination drug treatment of heart failure
  Arms: YanXinShi group
Drug: Trimetazidine pills — participants will take 20mg Trimetazidine pills TID in addition to the optimal combination drug treatment of heart failure
  Arms: Trimetazidine group
Drug: YanXinShi and Trimetazidine pills — participants will take 1800 mg YXS and 20 mg Trimetazidine pills TID in addition to the optimal combination drug treatment of heart failure
  Arms: YangXinShi and Trimetazidine group

SUMMARY:
The investigators set out to evaluate the effects of the traditional Chinese medicinal mixture under the brand name YangXinShi (YXS) on the prognosis in patients with chronic heart failure when it is combined with the optimal combination drug treatment of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* patients newly diagnosed with heart failure or have been diagnosed with chronic heart failure
* patients classified as NYHA II-IV (New York Heart Association)

Exclusion Criteria:

* with severe liver or renal dysfunction
* with severe systematic conditions such as infection, malignant hypertension etc.
* hemodynamic instability (arrhythmia, acute cardiac infarction, aortic dissection etc.)
* not cooperating due to psychomotor deficiency, or with contraindications for exercise testing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
change in EQ-5D Questionnaire | from baseline to 6 months
  health status measured in therms of five dimensions with the 5-level scale from 1-5, corresponding to having no problems and having extreme problems
change in EQ-VAS | from baseline to 6 months
  visual analogue scale (VAS) of EQ-5D Questionnaire scaled from 0-100, corresponding to the worse and the best health imagined

SECONDARY OUTCOMES:
change in disease specific quality of life | from baseline to 6 months
  assessment of disease-related QoL using Kansas City Cardiomyopathy Questionnaire (KCCQ-12) with 7 heart failure domains. Scores of each domain are scaled from 0-100, with 0 corresponding to the worst, 100 the best status.
change in heart rate variability | from baseline to 6 months
  assessed by Holter monitoring
change in left ventricular end-systolic diameters (in millimeters) | from baseline to 6 months
  assessed by echocardiographic examination
change in left ventricular end-diastolic diameters (in millimeters) | from baseline to 6 months
  assessed by echocardiographic examination
change in left ventricular ejection fraction (in percentage) | from baseline to 6 months
  assessed by echocardiographic examination
change in exercise tolerance | from baseline to 6 months
  assessed by the distance (in meters) walked on 6-minute walk test
change in metabolic equivalents (METs) | from baseline to 6 months
  measured as (volume of O2 (ml) consumption/kg/min) / (3.5 ml VO2/kg/min)
change in plasma N-terminal pro-B-type natriuretic peptide (NT-proBNP) levels (in pg/ml) | from baseline to 6 months
  assessed by blood tests

CONTACTS AND LOCATIONS:
Overall Officials: qin yu, M.D., Ph.D., Principal Investigator — Affiliated Zhongshan Hospital of Dalian University
Locations (1):
- Dept. of Cardiology, Affiliated Zhongshan hospital of Dalian University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided
age, gender, NYHA classification